CLINICAL TRIAL: NCT07217041
Title: A Pilot Clinical Study to Assess the Correlation Between Fluid Removal During Dialysis and HemoCept Device Data
Brief Title: Fluid Status of Dialysis Subjects
Status: Completed | Type: Observational
Sponsor: HemoCept Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRT-010
Record Dates: First submitted 2025-09-16; First posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: ESRD (End Stage Renal Disease)
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this clinical pilot study is to evaluate the ability of the device to properly detect the hydration status of the subject through the study of fluid removal data during dialysis and HemoCept device data.

ELIGIBILITY:
Inclusion Criteria:

* Study or representatives must have voluntarily signed the informed consent form before any study related procedures
* Subjects can be any gender, but must be between (and including) 18 and 75 years of age
* Subject has been on dialysis for more than 90 days and has been diagnosed with end stage kidney disease
* Subject is willing and able to provide informed consent and HIPAA authorization • Subject is able and willing to meet all study requirements
* Subject is able to place electrodes on bilateral deltoids and above the pant line on the waist

Exclusion Criteria:

* Subject is pregnant, breast-feeding, or intends to become pregnant during the course of the study.
* Subject has a personal medical history that includes:

  * Long Q-T syndrome
  * Cardiac channelopathies, genetic heart defects
  * Seizures
  * Acute untreated blood clotting disorders or acute untreated bleeding disorders
* Subject has had a heart transplant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects between (and including) the ages of 18 and 75 and who meet all the Inclusion/Exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Correlation between HemoCept device and changes in dry weight. | At specified points during dialysis treatment for 9 dialysis sessions, over the course of 3 weeks.
  The primary end point will be to determine if there is a correlation between HemoCept device data and dry weight changes during dialysis. The primary analysis will be conducted at specific points during dialysis treatment: prior to dialysis, in the middle of the dialysis session, and immediately following the completion of dialysis treatment.

SECONDARY OUTCOMES:
Device-related adverse events: device-related adverse events included all adverse events classified as definitely, probably, possibly, or undetermined relation to the device or procedure | From enrollment until the completion of 9 dialysis sessions, over a period of 3 weeks.
  All secondary endpoints will be summarized descriptively, and no hypothesis tests are planned.

CONTACTS AND LOCATIONS:
Locations (1):
- Sierra Nevad Specialty Care, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available